CLINICAL TRIAL: NCT06141382
Title: Development of Sensory Based Narrative Intervention and the Effect of Treatment on Vocabulary Development in Children - Pilot Study
Brief Title: Development of Sensory Based Narrative Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIPHAH/RCRS/REC/Letter-01202
Record Dates: First submitted 2023-11-09; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum disorder; Language disorders in children; Narrative therapy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- English Language-Sensory based narrative intervention (Experimental): This experimental group participants will receive sensory based intervention in English language.
  Interventions: Other: English Langugae-Sensory based narrative intervention
- English Language-Narrative intervention (Active Comparator): This Control group participants will receive narrative intervention in English language.
  Interventions: Other: English Language-Narrative intervention
- Urdu Language-Sensory based narrative intervention (Experimental): This experimental group participants will receive sensory based narrative intervention in Urdu language.
  Interventions: Other: Urdu Langusge-Sensory based narrative intervention
- Urdu Language-Narrative intervention (Active Comparator): This control group participants will receive narrative intervention in Urdu language.
  Interventions: Other: Urdu Language-Narrative intervention
- Bilingual-Sensory based narrative intervention (Experimental): This experimental group participants will receive sensory based narrative intervention in both English and Urdu language.
  Interventions: Other: Bilingual-Sensory based narrative intervention
- Bilingual-Narrative intervention (Active Comparator): This control group participants will receive narrative intervention in both English and Urdu language.
  Interventions: Other: Bilingual-Narrative intervention

INTERVENTIONS:
Other: English Langugae-Sensory based narrative intervention — Sensory based narrative intervention (auditory, visual and tactile stimulations) in English language will be administered on children with autism spectrum disorder (ASD). Intervention will be administered thrice a week in 45-minute-long session for 6 weeks.
  Arms: English Language-Sensory based narrative intervention
Other: English Language-Narrative intervention — Narrative intervention with the help of only pictures in English language will be administered on children with autism spectrum disorder (ASD). Intervention will be administred thrice a week in 45-minute long session for 6 weeks.
  Arms: English Language-Narrative intervention
Other: Urdu Langusge-Sensory based narrative intervention — Sensory based narrative intervention (auditory, visual and tactile stimulations) in Urdu language will be administered on children with autism spectrum disorder (ASD). Intervention will be administered thrice a week in 45-minute-long session for 6 weeks.
  Arms: Urdu Language-Sensory based narrative intervention
Other: Urdu Language-Narrative intervention — Narrative intervention with the help of only pictures in Urdu language will be administered on children with autism spectrum disorder (ASD). Intervention will be administered thrice a week in 45-minute long session for 6 weeks.
  Arms: Urdu Language-Narrative intervention
Other: Bilingual-Sensory based narrative intervention — Sensory based narrative intervention (auditory, visual and tactile stimulations) in both English and Urdu language will be administered on children with autism spectrum disorder (ASD). Intervention will be administered thrice a week in 45-minute-long session for 6 weeks.
  Arms: Bilingual-Sensory based narrative intervention
Other: Bilingual-Narrative intervention — Narrative intervention with the help of only pictures in both English and Urdu language will be administered on children with autism spectrum disorder (ASD). Intervention will be administered thrice a week in 45-minute long session for 6 weeks.
  Arms: Bilingual-Narrative intervention

SUMMARY:
The goal of this study is to develop a sensory based narrative intervention and see its effect on vocabulary development in children with autism spectrum disorder. Sensory based narrative intervention will be developed, and participants of experimental group will be given this treatment for 6 weeks. Control group participants will be given only narrative intervention. Vocabulary improvement will be documented pre-post testing in both groups.

DETAILED DESCRIPTION:
The present study aims to bridge an existing gap in the literature in Pakistan, as there are no evidence based therapeutic intervention tools available for narratives in Urdu.

The study further aims to provide a interventional resource pack for bilingual population who has Urdu as their first and dominant language. There is no therapeutic tool available for intervention that has incorporated multimodal sensory input for language intervention. Since tools developed internationally and from other countries cannot be incorporated due to cultural sensitivity and linguistic complexity, therefore, the current study will be able to incorporate these limitations. This study will provide a novel resource for intervention in the context of Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Participants with mild to moderate ASD aged between 6-11 years as assessed by ADOS (already diagnosed).
* CARS score 30-37 (mild to moderate)
* Both male and female participants.
* ASD participants at 2 Information Carrying word-level receptively and at Blank level 1 expressively. (will incorporate nouns, verbs and adjectives as per individual linguistic level).
* Participants with Urdu as their first language (home language) and English as a second language.

Exclusion Criteria:

* Individuals with any co-morbidity with Autism spectrum Disorder, such as hearing impairment, cleft lip and palate, visual impairment etc.
* Individuals with a mild to moderate diagnosis but severe behavioral difficulties
* Participants with any known sensory difficulties restricting use of certain sensory props.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 26 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Attention span | 18 days
  Changes from baseline, change in attention span will be measured in time in seconds pre and post intervention.
Sequencing skill | 18 days
  Change from baseline, sequencing skill will be measured as an ability to to place correct 3 part sequence picture of the story.
Vocabulary development | 18 days
  Change from baseline, vocabulary development will be measured through comprehension of individual grammatical categories such as nouns, verbs, adjectives and preposition pre and post frequency will be recorded through a record form and calculated.
Initiation for expression | 18 days
  change from baseline, initiation for expression will be documented in terms of time taken to initiate attempts at production level. It will be recorded on a record form with the help of stop watch on a record form.
Non verbal communication | 18 days
  change from baseline, non verbal communication attempts will be documented on a record form on each enlisted vocabulary word as highlighted by the blind reviewer pre and post testing.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Zubair, MS-SLP/T, Principal Investigator — Riphah International University
Locations (1):
- Profiles Speech & Language Therapy Clinic, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beatty J. What are narratives good for? Stud Hist Philos Biol Biomed Sci. 2016 Aug;58:33-40. doi: 10.1016/j.shpsc.2015.12.016. Epub 2016 Jan 21. PMID 26806602
- [Background] Barnes JL, Baron-Cohen S. The big picture: storytelling ability in adults with autism spectrum conditions. J Autism Dev Disord. 2012 Aug;42(8):1557-65. doi: 10.1007/s10803-011-1388-5. PMID 22042307
- [Background] Ferretti F, Adornetti I, Chiera A, Nicchiarelli S, Valeri G, Magni R, Vicari S, Marini A. Time and Narrative: An Investigation of Storytelling Abilities in Children With Autism Spectrum Disorder. Front Psychol. 2018 Jun 19;9:944. doi: 10.3389/fpsyg.2018.00944. eCollection 2018. PMID 29971024
- [Background] Ketelaars MP, Jansonius K, Cuperus J, Verhoeven L. Narrative competence in children with pragmatic language impairment: a longitudinal study. Int J Lang Commun Disord. 2016 Mar;51(2):162-73. doi: 10.1111/1460-6984.12195. Epub 2015 Nov 16. PMID 26935766
- [Background] Beytollahi S, Soleymani Z, Jalaie S. The Development of a New Test for Consecutive Assessment of Narrative Skills in Iranian School-Age Children. Iran J Med Sci. 2020 Nov;45(6):425-433. doi: 10.30476/ijms.2019.81984. PMID 33281259
- [Background] Venkatraman K, Thiruvalluvan V. Development of narratives in Tamil-speaking preschool children: A task comparison study. Heliyon. 2021 Jul 21;7(7):e07641. doi: 10.1016/j.heliyon.2021.e07641. eCollection 2021 Jul. PMID 34368487
- [Background] Abdalla F, Mahfoudhi A, Alhudhainah S. Structural Development of Narratives in Arabic: Task Complexity, Age, and Cultural Factors. Lang Speech Hear Serv Sch. 2020 Apr 7;51(2):405-415. doi: 10.1044/2019_LSHSS-19-00044. Epub 2020 Feb 20. PMID 32084324
- [Background] Bowles RP, Justice LM, Khan KS, Piasta SB, Skibbe LE, Foster TD. Development of the Narrative Assessment Protocol-2: A Tool for Examining Young Children's Narrative Skill. Lang Speech Hear Serv Sch. 2020 Apr 7;51(2):390-404. doi: 10.1044/2019_LSHSS-19-00038. Epub 2020 Feb 5. PMID 32073376